CLINICAL TRIAL: NCT06086860
Title: Effects of Mulligan Mobilization With and Without Dry Needling in Runner's Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0137 Mahnoor
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Runner's Knee
Keywords: Dry needling; Pain; Range of motion
MeSH Terms: conditions — Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan mobilization with dry needling. (Experimental): Participants in this group will receive Mulligan mobilization with dry needling.
  Interventions: Other: Mulligan mobilization with dry needling.
- Mulligan mobilization without dry needling. (Active Comparator): Participants in this group will receive Mulligan mobilization without dry needling.
  Interventions: Other: Mulligan mobilization without dry needling

INTERVENTIONS:
Other: Mulligan mobilization with dry needling. — The duration of intervention will be 6 weeks, 2 sessions a week, a total of 12 sessions will be given to the study participants. Each session will last for 30 minutes.
  Arms: Mulligan mobilization with dry needling.
Other: Mulligan mobilization without dry needling — The duration of intervention will be 6 weeks, 2 sessions a week, a total of 12 sessions will be given to the study participants. Each session will last for 30 minutes.
  Arms: Mulligan mobilization without dry needling.

SUMMARY:
The aim of this study is to determine the effects of Mulligan mobilization with and without dry needling on pain, range of motion, flexibility, functional disability and muscle strength in patients with Runner's Knee.

DETAILED DESCRIPTION:
Runner's knee or patellofemoral pain syndrome (PFPS) is a common cause of anterior knee pain in young active individuals. Patellofemoral pain (PFP), or anterior knee pain (AKP), is a common musculoskeletal disorder. It involves dysfunction in mechanical forces between the patella and the femur. The worldwide PFP prevalence has been reported as 15-45% of population. Females are at two times higher risk of PFP than males, especially young active females. The aim of this study is to determine the effects of Mulligan mobilization with and without dry needling in Runner's Knee in a randomized clinical trial.

The study will be randomized clinical trial. The study will be conducted at Johar Pain Relief Center, Lahore. The study will be completed within eight months after synopsis approval from ethical committee of Riphah College of Rehabilitation and Allied Health sciences. Sample size will be 40 (20 in each group). Non-probability convenience sampling technique will be used to recruit the Runner's Knee patients in the study and then they will be divided into two groups by simple randomization through sealed opaque envelope. Mulligan mobilization with dry needling will be given to group A. Mulligan mobilization without dry needling will be given to group B. Outcome measures will be pain, knee range of motion, flexibility, functional disability and muscle strength measured through Numeric pain rating scale (NPRS), goniometer, Kujala Patellofemoral Scale and Modified Sphygmomanometer Test (MST) respectively. Data will be analyzed by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders.
* Individuals aged 20-45 years with a clinical diagnosis of Runner's Knee.
* Participants experiencing retropatellar or anterior knee pain during at least two activities such as ascending and descending stairs, squatting, kneeling, or prolonged sitting, jumping or running.
* Pain scoring rate on numeric pain rating scale (NPRS) ≥ 3 during at least two activities.
* Duration lasting longer than two months.

Exclusion Criteria:

* Patients with a history of meniscus tears, bursitis, patellar tendon injury, ligamentous injury, joint degeneration, patellofemoral dislocation and / or recurrent subluxation.
* Participants with a history of arthritis.
* Individuals with a history of lower extremity surgery.
* Patients having knee pain referred from hip, lumbar spine and ankle joints.
* Any systemic disease and/or connective tissue disorders, or lumbosacral nerve root compression.
* Patients taking any pain medications.
* Individuals who previously received acupuncture therapy, injection, or dry needling technique for knee extensor muscle in last six months.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Pain: Numeric Pain Rating Scale (NPRS) | 6th Week
  Patients' overall assessment of pain will be provided using the numeric pain rating scale (NPRS). The NPRS is known to be a sensitive and reliable scale for clinical and experimental evaluation of pain intensity. The score ranges from 0, indicating no pain, to 10, expressing worst imaginable pain. The reliability of numeric pain rating scale (NPRS) is 0.92 (0.87, 0.95).
Functional Disability: Kujala Patellofemoral Scale (KPS) | 6th Week
  The Kujala score will be used to evaluate functional disability in patients with patellofemoral disorder. Kujala Patellofemoral Scale (KPS) is a 13-item, self completed instrument with different categories consisted of limping, weight bearing, walking, stairs, squatting, running, jumping, prolonged sitting, pain, swelling, painful patellar movements, muscle atrophy and flexion deficiency. The total score ranges from 0 to 100, with higher scores indicating lower levels of pain/ disability. It has been claimed that this tool is user-friendly and the test-retest reliability is highly acceptable. This tool is valid and sensitive for research purposes. The test-retest reliability is excellent with an intra-class correlation coefficient of 0.908 (p < 0.001; 95% CI [0.842-0.947]). The internal consistency is strong with Cronbach's alpha of 0.952 (p < 0.001).
Knee Range of Motion (ROM) (Flexion) : Goniometer | 6th Week
  Universal Goniometer is the most commonly utilised clinical tool for measuring joint range of motion due to its ease of use, low cost, and demonstrated reasonable levels of reliability and validity in numerous studies. Validity and intertester reliability (r =.97-.98; ICC =.98-.99) are both high.
Knee Range of Motion (ROM) (Extension) : Goniometer | 6th Week
  Universal Goniometer is the most commonly utilised clinical tool for measuring joint range of motion due to its ease of use, low cost, and demonstrated reasonable levels of reliability and validity in numerous studies. Validity and intertester reliability (r =.97-.98; ICC =.98-.99) are both high.
Flexibility: Goniometer | 6th Week
  Universal goniometer or inclinometer will be used for evaluating the knee joint range of motion and hamstring flexibility.
Muscle strength: Modified Sphygmomanometer Test (MST) | 6th Week
  A sphygmomanometer will be used for the evaluation of all muscular groups. A statistically significant correlation of moderate to high magnitude (0.58 ≤ r ≤ 0.81) is observed for concurrent validity of the MST with fixed stabilization for all muscle groups. Regarding inter-rater reliability, it is observed statistically significant ICC considered excellent to good (0.72 ≤ r ≤ 0.94) for all muscle groups. Regarding test-retest reliability, is good to excellent ICC (0.64 ≤ r ≤ 0.94) for all muscle groups. The MST with fixed stabilization is valid and reliable for clinical measurement of muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, Phd, Principal Investigator — Riphah International University
Locations (1):
- Johar Pain Relief Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rehman M, Riaz H. Comparison of mobilization with movement and Mulligan knee taping on Patellofemoral pain syndrome. J Pak Med Assoc. 2021 Sep;71(9):2119-2123. doi: 10.47391/JPMA.04-658. PMID 34580498
- [Background] Demirci S, Kinikli GI, Callaghan MJ, Tunay VB. Comparison of short-term effects of mobilization with movement and Kinesiotaping on pain, function and balance in patellofemoral pain. Acta Orthop Traumatol Turc. 2017 Dec;51(6):442-447. doi: 10.1016/j.aott.2017.09.005. Epub 2017 Oct 17. PMID 29054803
- [Background] Behrangrad S, Abbaszadeh-Amirdehi M, Kordi Yoosefinejad A, Esmaeilnejadganji SM. Comparison of dry needling and ischaemic compression techniques on pain and function in patients with patellofemoral pain syndrome: a randomised clinical trial. Acupunct Med. 2020 Dec;38(6):371-379. doi: 10.1177/0964528420912253. Epub 2020 Apr 27. PMID 32338532
- [Background] Sutlive TG, Golden A, King K, Morris WB, Morrison JE, Moore JH, Koppenhaver S. SHORT-TERM EFFECTS OF TRIGGER POINT DRY NEEDLING ON PAIN AND DISABILITY IN SUBJECTS WITH PATELLOFEMORAL PAIN SYNDROME. Int J Sports Phys Ther. 2018 Jun;13(3):462-473. PMID 30038832
- [Background] Espi-Lopez GV, Serra-Ano P, Vicent-Ferrando J, Sanchez-Moreno-Giner M, Arias-Buria JL, Cleland J, Fernandez-de-Las-Penas C. Effectiveness of Inclusion of Dry Needling in a Multimodal Therapy Program for Patellofemoral Pain: A Randomized Parallel-Group Trial. J Orthop Sports Phys Ther. 2017 Jun;47(6):392-401. doi: 10.2519/jospt.2017.7389. Epub 2017 May 13. PMID 28504067
- [Background] Ma YT, Li LH, Han Q, Wang XL, Jia PY, Huang QM, Zheng YJ. Effects of Trigger Point Dry Needling on Neuromuscular Performance and Pain of Individuals Affected by Patellofemoral Pain: A Randomized Controlled Trial. J Pain Res. 2020 Jul 7;13:1677-1686. doi: 10.2147/JPR.S240376. eCollection 2020. PMID 32753943
- [Background] Plummer S, Leonard J. Mobilization With Movement as Therapy to Reduce Knee Pain and Increase Knee Range of Motion. J Sport Rehabil. 2022 Jun 20;31(7):950-953. doi: 10.1123/jsr.2021-0294. Print 2022 Sep 1. PMID 35728804
- [Background] Freedman SR, Brody LT, Rosenthal M, Wise JC. Short-term effects of patellar kinesio taping on pain and hop function in patients with patellofemoral pain syndrome. Sports Health. 2014 Jul;6(4):294-300. doi: 10.1177/1941738114537793. PMID 24982700
- [Background] da Silva Boitrago MV, de Mello NN, Barin FR, Junior PL, de Souza Borges JH, Oliveira M. Effects of proprioceptive exercises and strengthening on pain and functionality for patellofemoral pain syndrome in women: A randomized controlled trial. J Clin Orthop Trauma. 2021 Apr 19;18:94-99. doi: 10.1016/j.jcot.2021.04.017. eCollection 2021 Jul. PMID 33996453
- [Background] da Cunha RA, Costa LO, Hespanhol Junior LC, Pires RS, Kujala UM, Lopes AD. Translation, cross-cultural adaptation, and clinimetric testing of instruments used to assess patients with patellofemoral pain syndrome in the Brazilian population. J Orthop Sports Phys Ther. 2013 May;43(5):332-9. doi: 10.2519/jospt.2013.4228. Epub 2013 Mar 13. PMID 23485881
- [Background] Mustamsir E, Phatama KY, Pratianto A, Pradana AS, Sukmajaya WP, Pandiangan RAH, Abduh M, Hidayat M. Validity and Reliability of the Indonesian Version of the Kujala Score for Patients With Patellofemoral Pain Syndrome. Orthop J Sports Med. 2020 May 28;8(5):2325967120922943. doi: 10.1177/2325967120922943. eCollection 2020 May. PMID 32523969
- [Background] Negahban H, Pouretezad M, Yazdi MJ, Sohani SM, Mazaheri M, Salavati M, Aryan N, Salehi R. Persian translation and validation of the Kujala Patellofemoral Scale in patients with patellofemoral pain syndrome. Disabil Rehabil. 2012;34(26):2259-63. doi: 10.3109/09638288.2012.683480. Epub 2012 May 27. PMID 22630589
- [Background] Apivatgaroon A, Angthong C, Sanguanjit P, Chernchujit B. The validity and reliability of the Thai version of the Kujala score for patients with patellofemoral pain syndrome. Disabil Rehabil. 2016 Oct;38(21):2161-4. doi: 10.3109/09638288.2015.1114035. Epub 2016 Jan 5. PMID 26729626
- [Background] Keogh JWL, Cox A, Anderson S, Liew B, Olsen A, Schram B, Furness J. Reliability and validity of clinically accessible smartphone applications to measure joint range of motion: A systematic review. PLoS One. 2019 May 8;14(5):e0215806. doi: 10.1371/journal.pone.0215806. eCollection 2019. PMID 31067247
- [Background] Pua YH, Poon CL, Seah FJ, Thumboo J, Clark RA, Tan MH, Chong HC, Tan JW, Chew ES, Yeo SJ. Predicting individual knee range of motion, knee pain, and walking limitation outcomes following total knee arthroplasty. Acta Orthop. 2019 Apr;90(2):179-186. doi: 10.1080/17453674.2018.1560647. PMID 30973090
- [Background] Souza LA, Martins JC, Moura JB, Teixeira-Salmela LF, De Paula FV, Faria CD. Assessment of muscular strength with the modified sphygmomanometer test: what is the best method and source of outcome values? Braz J Phys Ther. 2014 Mar-Apr;18(2):191-200. doi: 10.1590/s1413-35552012005000149. PMID 24839045
- [Background] Silva BBC, Venturato ACT, Aguiar LT, Filho LFRM, Faria CDCM, Polese JC. Validity and reliability of the Modified Sphygmomanometer Test with fixed stabilization for clinical measurement of muscle strength. J Bodyw Mov Ther. 2019 Oct;23(4):844-849. doi: 10.1016/j.jbmt.2019.05.008. Epub 2019 May 14. PMID 31733770